CLINICAL TRIAL: NCT02693028
Title: Lactobacillus Reuteri Feasibility Study on Probiotic Lozenges, Probiotic Chewing Gum and Probiotic Capsules and Perinatal Microbiome Seeding During Pregnancy
Brief Title: Lactobacillus Reuteri Feasibility Study on Probiotic Treatment and Perinatal Microbiome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Collaborators: BioGaia AB (Industry)
Responsible Party: Principal Investigator, Bo Jacobsson, Clinical professor, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Dnr. 085-15
Record Dates: First submitted 2015-10-12; First posted 2016-02-26 (Estimated); Last update posted 2018-12-12 (Actual); Status verified 2018-12

CONDITIONS: Pregnancy
Keywords: Microbiome; probiotic
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- probiotic lozenge (Active Comparator): Two probiotic lozenges per day (morning and evening) after meals. Enrollment will be done in gestational week 28-36. The treatment will last for the rest of pregnancy and six weeks post partum.
  Interventions: Drug: Probiotic lozenges
- Probiotic capsule (Active Comparator): Two probiotic capsules per day (morning and evening) after meals. Enrollment will be done in gestational week 28-36. The treatment will last for the rest of pregnancy and six weeks post partum.
  Interventions: Drug: Probiotic capsules
- Probiotic chewing gum (Active Comparator): The probiotic chewing gum should be chewed on for about 10 minutes. Enrollment will be done in gestational week 28-36. The treatment will last for the rest of pregnancy and six weeks post partum.
  Interventions: Drug: Probiotic chewing gum
- Placebo lozenge (Placebo Comparator): Two placebo lozenges per day (morning and evening) after meals. Enrollment will be done in gestational week 28-36. The treatment will last for the rest of pregnancy and six weeks post partum.
  Interventions: Drug: Placebo lozenges
- Placebo capsule (Placebo Comparator): Two placebo capsules per day (morning and evening) after meals. Enrollment will be done in gestational week 28-36. The treatment will last for the rest of pregnancy and six weeks post partum.
  Interventions: Drug: Placebo capsules

INTERVENTIONS:
Drug: Probiotic lozenges — The women participating in the study will take two probiotic lozenges per day (morning and evening) after meals.Enrollment will be done in gestational week 28-36. The treatment will last for the rest of pregnancy and six weeks post partum.
  Other Names: Lactobacillus reuteri lozenges
  Arms: probiotic lozenge
Drug: Placebo lozenges — The women participating in the study will take two placebo lozenges per day (morning and evening) after meals. Enrollment will be done in gestational week 28-36. The treatment will last for the rest of pregnancy and six weeks post partum.
  Other Names: "non active" treatment lozenges
  Arms: Placebo lozenge
Drug: Probiotic capsules — The women participating in the study will take two probiotic capsules per day (morning and evening) after meals. Enrollment will be done in gestational week 28-36. The treatment will last for the rest of pregnancy and six weeks post partum.
  Other Names: Lactobacillus reuteri capsules
  Arms: Probiotic capsule
Drug: Placebo capsules — The women participating in the study will take two placebo capsules per day (morning and evening) after meals. Enrollment will be done in gestational week 28-36. The treatment will last for the rest of pregnancy and six weeks post partum.
  Other Names: "non active" treatment capsules
  Arms: Placebo capsule
Drug: Probiotic chewing gum — The women participating in the study will take two probiotic chewing gums per day (morning and evening) after meals. Enrollment will be done in gestational week 28-36. The treatment will last for the rest of pregnancy and six weeks post partum.
  Other Names: Lactobacillus reuteri chewing gum
  Arms: Probiotic chewing gum

SUMMARY:
Investigators want to investigate if the Lactobacillus Reuteri (probiotic bacteria) given to pregnant women can be found in different maternal compartments and in the first stool and oral swab collected immediately after birth of a newborn delivered by cesarean delivery. Investigators also want to explore if exposure to this Lactobacillus Reuteri alters the level of inflammation in different compartments of the mother and the infant.

DETAILED DESCRIPTION:
The purpose of this project is to better understand the following issues:

1. How does bacteria transmit from the mother to the fetus and placenta during pregnancy and to the infant during the first 2-6 weeks after birth?
2. Does colonization of the pregnant mother and fetus/Child occur? How and when?
3. Can orally given probiotic bacteria be found in the newborn 2-6 weeks after birth, and if so where?
4. How is bacteria transported from the mother's intestinal lumen to the Child/fetus gut?
5. What impact has these bacteria on the level of inflammation in maternal and fetal compartments, especially that normally seen in the intestine of all newborns?
6. What impact has these bacteria in the bowel on a normal intestinal flora establishment?

ELIGIBILITY:
Inclusion Criteria:

* Single or multiple gestation
* Maternal age > or = 18 y

Exclusion Criteria:

* Known structural or chromosomal fetal malformation or abnormality
* Occlusive placenta previa, placenta previa in the anterior wall of the uterus, suspicion of accreta/increta/percreta infiltration
* Unable to understand information about the study due to language or severe mental disease
* Known Hepatitis B, C, HIV
* Known immunosuppressive illness if they are under treatment
* Treatment with cytokine, methotrexate or immunosuppresses cytotoxics in the last 6 months before the study.
* Gastro-intestinal surgery including gastric bypass or huge intestinal resection.
* Anaphylactic shock
* Uterus malformation that occludes cervical Canal or uterus segment.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-11; Primary Completion 2018-01 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Presence of Lactobacillus reuteri in different compartments in the mother and the Child. | Mother: From weeks 28-36 of pregnancy until 6 weeks post partum. Child: from birth till 4 years old.
  Both cultivation techniques for the specific bacteria and metagenomic techniques will be used to be able to study both cultivable and non-cultivable bacteria.

SECONDARY OUTCOMES:
Levels of Toll-like receptor stimulated with Lactobacillus plantarum, Pseudomonas aeruginosa and LPS after probiotic treatment and after placebo in different maternal and neonatal compartments. | Mother: From weeks 28-36 of pregnancy until 6 weeks post partum. Child: from birth till 4 years old.
  To evaluate whether there are differences in Toll-like receptor stimulation with Lactobacillus plantarum, Pseudomonas aeruginosa and LPS in different compartments between women treated with probiotic and the placebo group
Levels of IL-6, IL-10, IL-1beta, MCP-1, IL-17, TNF-alfa after probiotic treatment and after placebo in different maternal and neonatal compartments. | Mother: From weeks 28-36 of pregnancy until 6 weeks post partum. Child: from birth till 4 years old.
  To evaluate whether there are differences in the levels of cytokines and chemokines in different compartments between women treated with probiotic and the placebo group

CONTACTS AND LOCATIONS:
Overall Officials: Bo Jacobsson, Professor, Principal Investigator — Göteborg University
Locations (1):
- Sahlgrenska University Hospital, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Yeganegi M, Leung CG, Martins A, Kim SO, Reid G, Challis JR, Bocking AD. Lactobacillus rhamnosus GR-1 stimulates colony-stimulating factor 3 (granulocyte) (CSF3) output in placental trophoblast cells in a fetal sex-dependent manner. Biol Reprod. 2011 Jan;84(1):18-25. doi: 10.1095/biolreprod.110.085167. Epub 2010 Sep 1. PMID 20811016
- [Result] Aagaard K, Ma J, Antony KM, Ganu R, Petrosino J, Versalovic J. The placenta harbors a unique microbiome. Sci Transl Med. 2014 May 21;6(237):237ra65. doi: 10.1126/scitranslmed.3008599. PMID 24848255
- [Result] Cobo T, Kacerovsky M, Palacio M, Hornychova H, Hougaard DM, Skogstrand K, Jacobsson B. Intra-amniotic inflammatory response in subgroups of women with preterm prelabor rupture of the membranes. PLoS One. 2012;7(8):e43677. doi: 10.1371/journal.pone.0043677. Epub 2012 Aug 20. PMID 22916296
- [Result] Goncalves LF, Chaiworapongsa T, Romero R. Intrauterine infection and prematurity. Ment Retard Dev Disabil Res Rev. 2002;8(1):3-13. doi: 10.1002/mrdd.10008. PMID 11921380
- [Result] Jimenez E, Fernandez L, Marin ML, Martin R, Odriozola JM, Nueno-Palop C, Narbad A, Olivares M, Xaus J, Rodriguez JM. Isolation of commensal bacteria from umbilical cord blood of healthy neonates born by cesarean section. Curr Microbiol. 2005 Oct;51(4):270-4. doi: 10.1007/s00284-005-0020-3. Epub 2005 Sep 20. PMID 16187156
- [Result] Jimenez E, Marin ML, Martin R, Odriozola JM, Olivares M, Xaus J, Fernandez L, Rodriguez JM. Is meconium from healthy newborns actually sterile? Res Microbiol. 2008 Apr;159(3):187-93. doi: 10.1016/j.resmic.2007.12.007. Epub 2008 Jan 11. PMID 18281199
- [Result] Myhre R, Brantsaeter AL, Myking S, Gjessing HK, Sengpiel V, Meltzer HM, Haugen M, Jacobsson B. Intake of probiotic food and risk of spontaneous preterm delivery. Am J Clin Nutr. 2011 Jan;93(1):151-7. doi: 10.3945/ajcn.110.004085. Epub 2010 Oct 27. PMID 20980489
- [Result] Brantsaeter AL, Myhre R, Haugen M, Myking S, Sengpiel V, Magnus P, Jacobsson B, Meltzer HM. Intake of probiotic food and risk of preeclampsia in primiparous women: the Norwegian Mother and Child Cohort Study. Am J Epidemiol. 2011 Oct 1;174(7):807-15. doi: 10.1093/aje/kwr168. Epub 2011 Aug 5. PMID 21821542
- [Result] Bertelsen RJ, Brantsaeter AL, Magnus MC, Haugen M, Myhre R, Jacobsson B, Longnecker MP, Meltzer HM, London SJ. Probiotic milk consumption in pregnancy and infancy and subsequent childhood allergic diseases. J Allergy Clin Immunol. 2014 Jan;133(1):165-71.e1-8. doi: 10.1016/j.jaci.2013.07.032. Epub 2013 Sep 10. PMID 24034345
- [Result] Yeganegi M, Watson CS, Martins A, Kim SO, Reid G, Challis JR, Bocking AD. Effect of Lactobacillus rhamnosus GR-1 supernatant and fetal sex on lipopolysaccharide-induced cytokine and prostaglandin-regulating enzymes in human placental trophoblast cells: implications for treatment of bacterial vaginosis and prevention of preterm labor. Am J Obstet Gynecol. 2009 May;200(5):532.e1-8. doi: 10.1016/j.ajog.2008.12.032. Epub 2009 Mar 14. PMID 19285652